CLINICAL TRIAL: NCT00729248
Title: The Differential Effects of 3 Different Immunosuppressive Agents, Tacrolimus Mycophenolate Mofetil and Sirolimus on the Generation of Tregs and DCregs in in Vitro MLR and T Cell Activation Assays
Brief Title: The Differential Effects of 3 Different Immunosuppressive
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: Astellas Pharma US, Inc. (Industry)
Responsible Party: Principal Investigator, Lorenzo Gallon, Study Principal Investigator, Northwestern University
Other Study IDs: KV-08-001
Record Dates: First submitted 2008-08-04; First posted 2008-08-07 (Estimated); Results first posted 2013-08-28 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-05

CONDITIONS: Immunosuppression; Kidney Transplantation
Keywords: Transplants; Kidney Transplantation; Immunosuppression; Assay; Graft Rejection

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — White Cells.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The study is a laboratory investigation comparing the regulatory effects of different immunosuppressive therapies in an in vitro human MLR assay of selecting specific immunosuppressive therapy to promote a regulatory profile and determining possibly newer accepted dosing and drug concentrations for agents most associated with this regulatory profile.

DETAILED DESCRIPTION:
Life-long immunosuppressive (IS) therapy is typically required in the great majority of organ transplants. Immunobiologically correct IS dosing, tapering to low levels and/or monotherapy could lower the incidence of complications related to IS and improve long term graft and patient survival. The current standard of IS care for liver transplant recipients are the calcineurin-inhibitors (CNIs) tacrolimus (TAC) and cyclosporine (CSA), although alternative IS drugs such as mycophenolate mofetil (MMF) and sirolimus (SRL) are available for use in select patients. This is also true for kidney, pancreas and heart transplant recipients, with TAC being favored in each case. The ideal IS agent is one that can be given at low levels such that both rejection and long term toxicity are minimized. Directly related to IS minimization might be the development of a regulatory, "tolerance profile", as assessed by ex vivo immunophenotyping and functional assays that might test these specific IS agents singly, in combination or even in sequence.

Human Tregs and DCregs can be more predominantly generated in the presence of one of three IS agents with different modes of action, i.e., TAC, MMF or SRL, and in different conditions of antigen presentation and alloimmune incompatibility.

This is a bench protocol studying the effects of TAC, MMF and SRL on pre operative living renal recipient donor pair.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of Age or Older
* Undergoing living donor renal transplant

Exclusion Criteria:

* No active infection or history of malignancy
* No HIV infection
* No Hepatitis C (HCV) infection
* No prior transplant (kidney or other organ)
* No chromic use of immunosuppressive therapy or history of autoimmune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Six to Twelve preoperative renal transplant living donor pairs.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2008-07; Primary Completion 2009-07 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Gallon, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruit donor/recipient renal transplant subjects for blood draw before renal transplant surgery. Peripheral mononuclear cells (PBMC) were isolated from the blood, and were cultured in the following combinations: Recipient PMBC + Donor PBMC + No drug Recipient PMBC + Donor PBMC + Tacrolimus (TAC) Recipient PMBC + Donor PBMC + Sirolimus (SRL)
Groups:
- Participants: 12 participants were recruited/consented for the study. 2 subjects (donor/recipient pair) were withdrawn from the study. Ten participants (5 donors, 5 recipients) had blood drawn before renal transplant surgery. Peripheral mononuclear cells (PBMC) were isolated from the blood, and were cultured in the following combination: Recipient PMBC + Donor PBMC + Sirolimus (SRL)
Period: Overall Study
Arm/Group | Participants
Started | 12
Completed | 10
Not Completed | 2
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants (6 donors, 6 recipients) had blood drawn before renal transplant surgery. Peripheral mononuclear cells (PBMC) were isolated from the blood, and were cultured in the following combination:
  Recipient PMBC + Donor PBMC + No drug Recipient PMBC + Donor PBMC + Tacrolimus (TAC) Recipient PMBC + Donor PBMC + Sirolimus (SRL)
Arm/Group | All Participants
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 47.08 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: CD4+CD25 High FOXP3+ Cell Levels in Mixed Lymphocyte Reactions (MLRs) of Renal Pre-transplant Recipients/Donors
Description: CD4+CD25 high FOXP3+ cell levels in mixed lymphocyte reactions (MLRs) of Renal Pre-transplant Recipients/Donors were measured in the presence of 1) No Drug/Control; 2) 0.05-0.2, 0.3-3 and > 5 ng/ml Tacrolimus (TAC); OR 3) 0.05-0.2, 0.3-3 and > 5 ng/ml Sirolimus (SRL). CD4+CD25 high FOXP3+ cell levels in the MLRs with TAC or SRL are expressed as the percentage of CD4+CD25 high FOXP3+ cell levels in the MLRs with no drug.
Time Frame: 3 months
Population: For each arm, blood samples from 5 donor/recipient pairs (i.e., 10 participants) were used.
Measure: Mean (Standard Deviation); unit: Percentage of Control Cells
Groups:
- MLRs in the Presence of TAC: All participants (5 donors, 5 recipients) had blood drawn before renal transplant surgery. Peripheral mononuclear cells (PBMC) were isolated from the blood, and were cultured in the following combination:
  REcipient PMBC + Donor PBMC + Tacrolimus (TAC)
- MLRs in the Presence of SRL: All participants (5 donors, 5 recipietns) had blood drawn before renal transplant surgery. Peripheral mononuclear cells (PBMC) were isolated from the blood, and were cultured in teh following combination:
  Recipient PMBC + Donor PBMC + Sirolimus (SRL)
Arm/Group | MLRs in the Presence of TAC | MLRs in the Presence of SRL
Number analyzed (Participants) | 10 | 10
Percentage of Control Cells
  Cell Levels in 0.05-0.2 ng/mL TAC or SRL | 90 (20) | 85 (5)
  Cell Levels in 0.3-3 ng/mL TAC or SRL | 25 (15) | 50 (10)
  Cell Levels in > 5 ng/mL TAC or SRL | 10 (5) | 45 (10)

ADVERSE EVENTS:
Groups:
- All Participants: All participants (6 donors, 6 recipients) had blood drawn before renal transplant surgery. Peripheral mononuclear cells (PBMC) were isolated from the blood, and were cultured in the following combination: Recipient PMBC + Donor PBMC + Sirolimus (SRL)
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No